CLINICAL TRIAL: NCT02721654
Title: Comparison of Plasmalyte 148® and Saline for Fluid Resuscitation and Intravenous Fluid Therapy in Critically Ill Adults
Brief Title: Plasma-Lyte 148® versUs Saline Study
Acronym: PLUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: Australian and New Zealand Intensive Care Society Clinical Trials Group (Network); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GI-CCT7587; U1111-1178-8334 (Other: World Health Organisation (WHO) Universal Trial Number (UTN))
Record Dates: First submitted 2016-03-15; First posted 2016-03-29 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Hypovolemia
Keywords: Plasma-Lyte; Sodium chloride; Saline; Fluid resuscitation; Intravenous fluid therapy; Critically ill; Critical care
MeSH Terms: conditions — Hypovolemia; Critical Illness | interventions — Plasma-lyte 148; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma-Lyte 148® (Experimental): Following randomisation, each study participant will receive either Plasma-Lyte 148® or 0.9% saline alone for all resuscitation episodes and for all compatible intravenous crystalloid therapy while in ICU (for up to 90 days).
  Interventions: Drug: Plasma-Lyte 148®
- 0.9% sodium chloride (Active Comparator): Following randomisation, each study participant will receive either Plasma-Lyte 148® or 0.9% saline alone for all resuscitation episodes and for all compatible intravenous crystalloid therapy while in ICU (for up to 90 days).
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: Plasma-Lyte 148® — Plasma-Lyte 148 (approx pH 7.4) IV infusion is a sterile, clear nonpyrogenic isotonic solution & when administered intravenously it is a source of water, electrolytes & calories. Plasma-Lyte 148 intravenous infusion is indicated as a source of water & electrolytes or as an alkalinising agent.
  Other Names: Balanced crystalloid solution
  Arms: Plasma-Lyte 148®
Drug: 0.9% sodium chloride — The active ingredient is sodium chloride formulated in Water for Injections. The chemical name is sodium chloride with molecular formula NaCl. Sodium Chloride (0.9%) intravenous infusion preparation is a sterile & non-pyrogenic solution & is indicated for extracellular fluid replacement & in the management of metabolic alkalosis in the presence of fluid loss, & for restoring or maintaining the concentration of sodium & chloride ions. As sodium chloride intravenous infusion is administered to the systemic circulation by intravenous infusion, the bioavailability (absorption) of the active components is complete (100 per cent).
  Other Names: Saline
  Arms: 0.9% sodium chloride

SUMMARY:
The aim of PLUS is to conduct a multi-centre, blinded, randomised, controlled trial (RCT) to determine whether fluid resuscitation and therapy with a "balanced" crystalloid solution (Plasma-Lyte 148®) decreases 90-day mortality in critically ill patients requiring fluid resuscitation when compared with the same treatment using 0.9% sodium chloride (saline)

DETAILED DESCRIPTION:
Fluid resuscitation is a fundamental component of the management of acutely and critically ill patients and the choice of fluid is a longstanding issue of debate.

Worldwide, 0.9% saline has traditionally been the most widely used resuscitation fluid, however its use is increasingly challenged by emerging evidence that suggests its high chloride content may have clinically important adverse effects and that resuscitation with so-called "balanced" or "buffered" crystalloids (such as Plasma-Lyte 148®) offer patients better outcomes.

Given the limitations of current evidence, there is now a scientific, ethical and health economic imperative to provide an accurate and reliable estimate of the comparative risks versus benefit of Plasma-Lyte 148® versus 0.9% saline.

The PLUS study is a prospective, multi-centre, parallel group, concealed, blinded, randomised, controlled trial.

The study will test the hypothesis that in a heterogeneous population of critically ill adults, random assignment to Plasma-Lyte 148® for intravascular volume resuscitation and crystalloid fluid therapy in the Intensive Care Unit (ICU) results in different 90-day all-cause mortality when compared with random assignment to 0.9% sodium chloride (saline) for the same treatment.

Each patient who meets all inclusion criteria and no exclusion criteria will be randomised to receive either Plasma-Lyte 148® or 0.9% saline for all resuscitation episodes and for all compatible crystalloid therapy while in ICU for up to 90 days after randomisation. Other crystalloid fluids may be used as carrier fluids for the infusion of any drug for which either Plasma-Lyte 148® or 0.9% saline is considered incompatible.The study treatments will be supplied in identical 1000 ml bags and treatment assignment will be concealed.

The volume of study fluid being administered will be titrated against clinical endpoints determined by the treating clinicians and reviewed as clinically appropriate during the period of resuscitation and ICU treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient will receive fluid resuscitation defined as a bolus of fluid, prescribed to be administered over one hour or less to increase or maintain intravascular volume that is in addition to maintenance fluids, or specific fluids used to replace non-physiological fluid losses
* The patient is expected to be in the ICU the day after tomorrow
* The patient is not expected to be well enough to be eating tomorrow
* An arterial or central venous catheter is in situ, or placement is imminent as part of routine management
* Both Plasma-Lyte 148® and 0.9% saline are considered equally appropriate for the patient
* The requirement for fluid resuscitation is supported by at least one of seven pre-specified clinical signs: heart rate > 90 beats per minute; systolic blood pressure < 100 mmHg or mean arterial pressure < 75 mmHg; central venous pressure < 10 mmHg; pulmonary artery wedge pressure < 12 mmHg; capillary refill time > 1 second; OR urine output < 0.5 ml/kg for at least one hour

Exclusion Criteria:

* Age less than 18 years
* Patients who have received more than 500mls of fluid resuscitation (as defined above) prescribed in the ICU during this current ICU admission
* Patients transferred directly from another ICU who have received more than 500mls of fluid resuscitation (as defined above) during that ICU admission
* Contraindication to either study fluid e.g. previous allergic reaction to Plasma-Lyte 148®
* Patients admitted to the ICU with specific fluid requirements: the treatment of burns; following liver transplantation surgery; for correction of specific electrolyte abnormalities
* Patients with traumatic brain injury or those considered at risk of developing cerebral oedema
* Patients in whom death is deemed imminent and inevitable
* Patients with an underlying disease process with a life expectancy of <90 days
* Patients in whom it is unlikely the primary outcome can be ascertained
* Patients who have previously been enrolled in PLUS
* Known or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5037 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Death from all causes | At 90 days after randomisation

SECONDARY OUTCOMES:
Mean and peak serum creatinine concentration | First seven days
ICU, hospital and 28 day all-cause mortality | 28 days and 6 months after randomisation
Duration of ICU stay | 28 days and 90 days after randomisation
Duration of Hospital stay | 28 days and 90 days after randomisation
Proportion of patients newly treated with renal replacement therapy | up to 90 days after randomisation.
Duration of mechanical ventilation in ICU | 90 days after randomisation
Proportion of patients treated with and duration of treatment with vasoactive drugs | 90 days after randomisation
Quality of life assessment using the EQ-5D-5L questionnaire | At 6 months after randomisation
Maximum post-randomisation increase in serum creatinine in ICU during the index hospital admission. | 90 days after randomisation
Healthcare services usage during the six months after randomisation by healthcare record linkage using state and national data linkage units | During the six months after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Simon Finfer, Professor, Study Chair — The George Institute
Locations (51):
- Australia (39):
  - Blacktown Hospital, Blacktown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - The Sutherland Hospital, Caringbah, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Hornsby Ku-ring-gai Hospital, Hornsby, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Nepean, Penrith, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Wagga Wagga Rural Referral Hospital, Wagga Wagga, New South Wales
  - The Sydney Adventist Hospital, Wahroonga, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - The Wesley Hospital, Auchenflower, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Robina Hospital, Robina, Queensland
  - Mater Misericordiae, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Ballarat Health Services, Ballarat, Victoria
  - Bendigo Hospital, Bendigo, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - Footscray Hospital, Western Health, Footscray, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Maroondah Hospital, Ringwood East, Victoria
  - Sunshine Hospital, Western Health, St Albans, Victoria
  - St John of God Murdoch Hospital, Murdoch, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
- New Zealand (12):
  - North Shore Hospital, Takapuna, Auckland
  - Rotorua Hospital, Rotorua, Bay of Plenty
  - Hawkes Bay, Hastings, Camberley
  - Christchurch Hospital, Christchurch, Canterbury
  - Hutt Hospital, Lower Hutt, Wellington Region
  - Wellington Hospital, Newtown, Wellington Region
  - Auckland City Hospital (CVICU), Auckland
  - Auckland City Hospital (DCCM), Auckland
  - Middlemore Hospital, Auckland
  - Waikato Hospital, Hamilton
  - Nelson Hospital, Nelson
  - Tauranga Hospital, Tauranga

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Finfer S, Micallef S, Hammond N, Navarra L, Bellomo R, Billot L, Delaney A, Gallagher M, Gattas D, Li Q, Mackle D, Mysore J, Saxena M, Taylor C, Young P, Myburgh J; PLUS Study Investigators and the Australian New Zealand Intensive Care Society Clinical Trials Group. Balanced Multielectrolyte Solution versus Saline in Critically Ill Adults. N Engl J Med. 2022 Mar 3;386(9):815-826. doi: 10.1056/NEJMoa2114464. Epub 2022 Jan 18. PMID 35041780